CLINICAL TRIAL: NCT03868410
Title: A Novel Approach for Brain Stimulation in Severe Stroke
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ela B. Plow, Assistant Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-861
Record Dates: First submitted 2018-09-24; First posted 2019-03-11 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: stroke; brain stimulation; TMS; Upper Limb; MRI; CVA; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: In a pilot, randomized, assessor-blind clinical trial, an anticipated 24 patients will be assigned to either receive stimulation to a new brain target- contralesional dorsal premotor cortex (cPMd) located in the non-stroke hemisphere- or the conventional brain target- ipsilesional primary motor cortex (iM1) located in the stroke hemisphere. Stimulation will be delivered in conjunction with rehabilitation for 2 days a week for 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: Subjects will be told they will receive brain stimulation, but will be given no indication as to which target will be stimulated. Investigators analyzing functional outcome data, neurophysiology data and MRI data will receive coded data that conceals the identity of the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Contralesional dorsal premotor cortex (cPMD) rTMS + Training (Active Comparator): New Approach
  Interventions: Device: New Repetitive Magnetic Stimulation (rTMS) Approach
- Ipsilesional Primary Motor Cortex (iM1) rTMS + Training (Active Comparator): Conventional Approach
  Interventions: Device: Conventional Repetitive Magnetic Stimulation (rTMS) Approach

INTERVENTIONS:
Device: New Repetitive Magnetic Stimulation (rTMS) Approach — Participants in this arm will receive rTMS-based facilitation of the contralesional dorsal premotor cortex (cPMd) located in the non-stroke hemisphere before start of each session. High-frequency rTMS (5-Hz) will be delivered using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
  Other Names: Contralesional dorsal premotor cortex (cPMD) rTMS + Training
  Arms: Contralesional dorsal premotor cortex (cPMD) rTMS + Training
Device: Conventional Repetitive Magnetic Stimulation (rTMS) Approach — Participants in this arm will receive rTMS-based facilitation of the ipsilesional primary motor cortex (iM1) before the start of each session. iM1 will be stimulated with high-frequency rTMS (5-Hz) using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
  Other Names: Ipsilesional Primary Motor Cortex (iM1) rTMS + Training
  Arms: Ipsilesional Primary Motor Cortex (iM1) rTMS + Training

SUMMARY:
The long-term goal of this project is to develop upper limb rehabilitation interventions that can be utilized for stroke survivors, specifically survivors with more severe limitations in use of their affected upper limb.

This study will utilize a novel method of non-invasive brain stimulation in conjunction with upper limb training given for 12 visits over a period of 6 weeks.

The study will include the following site visits:

* Eligibility Screening and Informed Consent Visit
* An MRI visit
* Two testing visits in which motor function of the upper limb and neurophysiology will be measured
* 12 intervention visits during which patients will receive upper limb training in conjunction with non-invasive brain stimulation
* Repeat testing of motor function of the upper limb and neurophysiology
* Repeat MRI testing
* A follow-up visit completed 3 months after the completion of interventions

DETAILED DESCRIPTION:
In a pilot, randomized clinical trial, 24 stroke patients with moderate/severe impairments will receive non-invasive brain stimulation (repetitive Transcranial Magnetic Stimulation or rTMS) to one of two targets in the brain in conjunction with upper limb training for 2 days a week for 6 weeks. The primary outcome will be upper limb motor impairment, and secondary outcomes will be tests of functional abilities, proximal motor control, and patient-reported disability. Associated neural mechanisms will also be studied using neurophysiological and functional connectivity MRI techniques. Damage to ipsilesional corticospinal pathways will be indexed with diffusion tensor imaging (DTI).

ELIGIBILITY:
Inclusion Criteria:

* chronic phase (≥6 months) after index stroke
* moderate or severely impaired (UEFM ≤42)
* have either extensive damage to ipsilesional pathways (MEP-), or, have one of the following: less than 10 degrees active wrist extension, less than 10 degrees active thumb extension/abduction, less than 10 degrees active extension in at least 2 additional digits (i.e. will not meet minimum Constraint-Induced Movement Therapy [CIMT] criteria).
* medically stable

Exclusion Criteria:

* cerebellar stroke
* brainstem stroke
* bilateral strokes affecting sensorimotor structures
* severe cognitive impairment
* substantially elevated tone/spasticity in wrist/hand (Modified Ashworth Scale >3)
* severe contracture
* participation in outpatient or Botox therapy within 2 months
* exclusion criteria for TMS and MRI (metal implant in head, H/O seizures, alcohol or substance abuse, intake of medications contraindicated with TMS, cardiac pacemaker or programmable implant).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ela Plow, PhD, Principal Investigator — Lerner Research Institute; Cleveland Clinic Foundation
Locations (1):
- Lerner Research Institute; Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham DA, Varnerin N, Machado A, Bonnett C, Janini D, Roelle S, Potter-Baker K, Sankarasubramanian V, Wang X, Yue G, Plow EB. Stimulation targeting higher motor areas in stroke rehabilitation: A proof-of-concept, randomized, double-blinded placebo-controlled study of effectiveness and underlying mechanisms. Restor Neurol Neurosci. 2015;33(6):911-26. doi: 10.3233/RNN-150574. PMID 26484700
- [Background] Potter-Baker KA, Lin YL, Machado AG, Conforto AB, Cunningham DA, Sankarasubramanian V, Sakaie K, Plow EB. Variability of motor evoked potentials in stroke explained by corticospinal pathway integrity. Brain Stimul. 2018 Jul-Aug;11(4):929-931. doi: 10.1016/j.brs.2018.03.004. Epub 2018 Mar 9. No abstract available. PMID 29563050
- [Background] Plow EB, Cunningham DA, Varnerin N, Machado A. Rethinking stimulation of the brain in stroke rehabilitation: why higher motor areas might be better alternatives for patients with greater impairments. Neuroscientist. 2015 Jun;21(3):225-40. doi: 10.1177/1073858414537381. Epub 2014 Jun 20. PMID 24951091
- [Result] Sankarasubramanian V, Machado AG, Conforto AB, Potter-Baker KA, Cunningham DA, Varnerin NM, Wang X, Sakaie K, Plow EB. Inhibition versus facilitation of contralesional motor cortices in stroke: Deriving a model to tailor brain stimulation. Clin Neurophysiol. 2017 Jun;128(6):892-902. doi: 10.1016/j.clinph.2017.03.030. Epub 2017 Mar 21. PMID 28402865
- [Derived] Li X, Lin YL, Cunningham DA, Wolf SL, Sakaie K, Conforto AB, Machado AG, Mohan A, O'Laughlin K, Wang X, Widina M, Plow EB. Repetitive Transcranial Magnetic Stimulation of the Contralesional Dorsal Premotor Cortex for Upper Extremity Motor Improvement in Severe Stroke: Study Protocol for a Pilot Randomized Clinical Trial. Cerebrovasc Dis. 2022;51(5):557-564. doi: 10.1159/000521514. Epub 2022 Jan 20. PMID 35051941

RESULTS

PARTICIPANT FLOW:
Groups:
- cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training: New Approach
  New rTMS Approach: Participants in this arm will receive rTMS-based facilitation of the contralesional dorsal premotor cortex (cPMd) located in the non-stroke hemisphere before start of each session. High-frequency rTMS (5-Hz) will be delivered using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
- iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training: Conventional Approach
  Conventional rTMS Approach: Participants in this arm will receive rTMS-based facilitation of the ipsilesional primary motor cortex (iM1) before the start of each session. iM1 will be stimulated with high-frequency rTMS (5-Hz) using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
Period: Overall Study
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Started | 8 | 8
Completed | 8 | 7
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adults with chronic (>6 months) unilateral upper limb motor deficits post-stroke.
Groups:
- Total: Total of all reporting groups
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (13.7) | 65.3 (10.1) | 64.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Stroke Type [Count of Participants; unit: Participants]
  hemorrhagic | 2 | 1 | 3
  ischemic | 6 | 7 | 13
Dominant Paresis [Count of Participants; unit: Participants]
  yes | 5 | 6 | 11
  no | 3 | 2 | 5
Active wrist extension [Count of Participants; unit: Participants]
  yes | 5 | 4 | 9
  no | 3 | 4 | 7
Resting Transcranial Magnetic Stimulation (TMS) Motor Evoked Potential (MEP) [Count of Participants; unit: Participants]
  yes | 2 | 2 | 4
  no | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Fugyl-Meyer Score (UEFM)
Description: Change between Baseline and Post-Test (average 6 weeks) is reported for the UEFM. Impairment will be measured using UEFM, one of the most widely used assessments in stroke. UEFM will serve as our primary outcome because it is sensitive to discerning the effects of rTMS/rehabilitation, and has excellent reliability (ICC= 0.97), consistency (Cronbach's α= 0.84) and validity. UEFM has a score ranging from 0-66 (0 meaning there is no movement of the paretic arm, and 66 meaning there is no functional limitation of the paretic arm.)
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: change score from baseline to post-test
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
change score from baseline to post-test | 2.625 (0.498) | 2.625 (0.680)

2. Primary Outcome: Change in Inter-hemispheric Inhibition (IHI)
Description: Inter-hemispheric connectivity (IHI) will be collected with transcranial magnetic stimulation (TMS) and is assessed using ipsilateral silent period (ISP) method. TMS is delivered to the contralesional motor hotspot at supra-maximal intensity (100% maximum stimulator output) while participants maintain sub-maximal contraction (50% maximum volitional contraction) of the ipsilateral paretic extensor digitorum communis muscle for 40 trials. Ipsilateral TMS produces transient suppression of on-going EMG activity, called ISP. ISP is analyzed using an algorithm that compares psotstimulus average rectified EMG to mean consecutive difference (MCD) of background EMG. A threshold of MCD x1.77 below mean background EMG is used to define ISP onset and offset. ISP duration is then calculated as a difference between onset and offset of the ISP.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
milliseconds | -8.8774 (4.62765) | 3.04521 (4.62765)

3. Secondary Outcome: Change in Wolf Motor Function Test (WMFT) Functional Ability
Description: Change in Functional Ability (FA) from Baseline to Post-Test (average 6 weeks) is reported for the Wolf Motor Function Test. Functional ability (FA) to use the paretic upper limb in a variety of tasks will be assessed using WMFT. FA is scored on a scale from 0-5 with 0 not attempting the task at all and 5 being completely normal movement compared to non paretic limb. 15 items of WMFT are given a FA for the Paretic limb and then the score is averaged to give an overall FA for each participant.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
units on a scale | 0.083 (0.047) | 0.217 (0.077)

4. Secondary Outcome: Change in Wolf Motor Function Test (WMFT) Rate Paretic Limb
Description: Change in Rate of the Paretic limb from Baseline to Post-Test (average 6 weeks) is reported for the Wolf Motor Function Test. Time to complete each task will be noted and converted to rate (60/Performance Time (sec)), optimized for measurement in moderately/severely-impaired patients. The rate will be calculated for the Paretic limb [WMFT Rate (P)]. The higher the rate the quicker they were able to complete the task.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: Tasks per minute
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
Tasks per minute | 0.970 (0.682) | 2.972 (1.165)

5. Secondary Outcome: Change in Wolf Motor Function Test (WMFT) Rate Non-paretic Limb
Description: Change in Rate of the Non-paretic limb from Baseline to Post-Test (average 6 weeks) is reported for the Wolf Motor Function Test. Time to complete each task will be noted and converted to rate (60/Performance Time (sec)), optimized for measurement in moderately/severely-impaired patients. The rate will be calculated for the Non-paretic limb [WMFT Rate (NP)]. The higher the rate the quicker they were able to complete the task.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: Tasks per minute
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
Tasks per minute | 2.552 (1.048) | 3.098 (0.977)

6. Secondary Outcome: Change in Wolf Motor Function Test (WMFT) Rate Paretic Limb Normalized to the Non-paretic Limb
Description: Change in the normalized Rate of the Paretic limb to the Non-paretic limb from Baseline to Post-Test (average 6 weeks) is reported for the Wolf Motor Function Test. Time to complete each task will be noted and converted to rate (60/Performance Time (sec)), optimized for measurement in moderately/severely-impaired patients. The rate will be calculated for the Paretic limb normalized to the Non-paretic limb [WMFT Rate (P/NP)]. The higher the rate the quicker they were able to complete the task.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: Tasks per minute
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
Tasks per minute | 1.593 (1.477) | 2.921 (1.306)

7. Secondary Outcome: Change in Stroke Impact Scale (SIS-16)
Description: Change in total score between Baseline and Post-Test (average 6 weeks) is reported for the Stoke Impact Scale (SIS-16) for each group. Patient's perceived disability related to physical function will be indexed using the Stroke Impact Scale (SIS-16) which a subjective questionnaire asked to the subject pertaining of 16 questions. Each question is rated on scale from 1 to 5 and then the scores are totaled. Total scores can range from 16-80 (16 means that none of the functional tasks asked can be performed, a score of 80 means the subject has no issues at all performing any of the tasks asked).
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | cPMD Repetitive Transcranial Magnetic Stimulation (rTMS) + Training | iM1 Repetitive Transcranial Magnetic Stimulation (rTMS) + Training
Number analyzed (Participants) | 8 | 7
score on a scale | 4.250 (1.264) | 1.375 (1.802)

8. Secondary Outcome: Change Resting State Functional Magnetic Resonance Imaging(rsfMRI)
Description: Functional connectivity will complement IHI measurement as a secondary outcome because while IHI records neurophysiologic interactions between a contralesional and a weak ipsilesional region, functional connectivity defines "global" interactions across multiple regions.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-04

9. Secondary Outcome: Change in Ipsilateral MEPs (Motor Evoked Potentials)
Description: Output of uncrossed pathways will be studied as ipsilateral MEPs elicited in the paretic-muscle with TMS.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-04

10. Secondary Outcome: Diffusion Tensor Imaging (DTI)
Description: Diffusion Tensor Imaging (DTI) enables the investigation of structural integrity and orientation of pathways in vivo through the estimation of magnitude and directionality of water diffusion. DTI metrics can help quantitate damage even when patients show no response to Transcranial Magnetic Stimulation (TMS) due to extensive damage (MEP-). Ipsilesional and contralesional corticospinal tracts will be reconstructed using probabilistic tractography. Fractional Anisotropy (FA), a unit-less measure of white matter integrity, will be calculated.
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-04

11. Secondary Outcome: Change in SULCS
Description: Change in total score between Baseline and Post-Test (average 6 weeks) is reported for the Stroke Upper Limb Capacity Scale (SULCS). SULCS is a stroke-specific assessment instrument that evaluates functional capacity of the upper limb based on the execution of 10 tasks. Score ranges from 0-10 where 0 is the lowest level of function in which the participant cannot perform any of the tasks as instructed and 10 is the highest level of function in which all 10 tasks are completed as instructed.
Time Frame: Change between Baseline and Post-Test (average 6 weeks)
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: Each participant was monitored from Baseline assessment through 3 month follow-up (~5.5 months)
Groups:
- cPMD rTMS + Training: New Approach
  New rTMS Approach: Participants in this arm will receive rTMS-based facilitation of the contralesional dorsal premotor cortex (cPMd) located in the non-stroke hemisphere before start of each session. High-frequency rTMS (5-Hz) will be delivered using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
- iM1 rTMS + Training: Conventional Approach
  Conventional rTMS Approach: Participants in this arm will receive rTMS-based facilitation of the ipsilesional primary motor cortex (iM1) before the start of each session. iM1 will be stimulated with high-frequency rTMS (5-Hz) using 42 10-sec trains of 50 pulses each (total 2100 pulses) for a period of 24 minutes. Immediately after the completion of rTMS, participants will undergo upper limb training for a total of one hour. Participants will receive these interventions 2 days a week for 6 weeks, i.e., for a total of 12 sessions.
Arm/Group | cPMD rTMS + Training | iM1 rTMS + Training
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cPMD rTMS + Training (N=8) | iM1 rTMS + Training (N=8)
headache (Nervous system disorders) | 1 (2) | 0 (0) — headache after receiving TMS
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — neck pain after receiving TMS
scalp irritation (Nervous system disorders) | 0 (0) | 1 (1) — scalp irritation after receiving TMS
dizziness/lightheaded (Nervous system disorders) | 1 (1) | 1 (1) — dizziness/lightheaded after receiving TMS
High Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1) — High Blood Pressure recorded during the session
Fall at home (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03868410/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03868410/SAP_001.pdf